CLINICAL TRIAL: NCT05090462
Title: The Use of PICO Dressings for Patients Undergoing Emergency Laparotomy
Brief Title: PICO Dressings for Emergency Laparotomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: North Middlesex University Hospital NHS Trust (Other Government)
Responsible Party: Principal Investigator, Nader Bedwani, Principal Investigator, North Middlesex University Hospital NHS Trust
Other Study IDs: 1234
Record Dates: First submitted 2021-10-08; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard surgical dressings (Clearpore)
- NPWT dressing (PICO)
  Interventions: Device: PICO dressing

INTERVENTIONS:
Device: PICO dressing — Negative Pressure Wound Therapy device
  Groups: NPWT dressing (PICO)

SUMMARY:
SSI (Surgical Site Infection) rate is an important consideration after emergency laparotomy. SSIs carry a high financial burden for health institutes with the cost of major SSIs after emergency laparotomy to add an additional cost of £10000-£15000 per patient.

NICE has recommended the use of PICO dressings for the reduction of SSI rate as a cost-neutral.

The purpose of this study was to review the current SSI rate, assess the patient risk factors for development of SSIs and evaluate if the use of PICO dressings as per NICE guidelines will reduce the SSI rate.

ELIGIBILITY:
Inclusion Criteria:

* All emergency midline laparotomy
* Laparoscopic converted open

Exclusion Criteria:

- Reoperation with 28 days of index laparotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients (>/= 18 years) undergoing emergency (laparotomy) surgery at a single centre (North Middlesex University Hospital, London, UK) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
SSI Day 7 | Day 7
  Presence of SSI

SECONDARY OUTCOMES:
SSI Day 7 | Day 28
  Presence of SSI
Length of stay | through study completion, an average of 6 months
  Length of stay
Surgical site complications | Day 28
  Number of participants with other complications of the wound to include dehiscence and burst abdomen
Reoperation | Day 28
  Number of participants undergoing reoperation
SSI grading | Day 28
  SSI grading as per Southampton scoring system (if applicable) (Grade 0-5 with 5 being worse outcome)
Length of antibiotic therapy | Day 28
  Duration of post-operative antibiotic therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Nader University Bedwani, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Will be shared through IRAS
Supporting Information: Study Protocol, SAP